CLINICAL TRIAL: NCT02007421
Title: The Natural History of Anal Human Papillomavirus Infection and Anal Cellular Abnormalities in Homosexual Men
Brief Title: Study of the Prevention of Anal Cancer
Acronym: SPANC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPANC; NHMRC (Other Grant/Funding Number: NRMRC)
Record Dates: First submitted 2013-11-26; First posted 2013-12-10 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Human Papillomavirus; Cancer
Keywords: Human Papillomavirus,; Anal High Grade Squamous intraepithelial lesions,; Homosexual Men; High resolution anoscopy,; Cancer Screening; HIV
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV positive homosexual men (Other): Therefore, it is proposed we conduct a longitudinal study of the epidemiology of low risk and high risk HPV infection and related low grade and high grade anal cancers in HIV negative and HIV positive homosexual men who are 35 years or older. Participants are asked questions about recent experiences of anal intercourse in the last six months.
  At baseline, all men (both HIV positive and HIV negative)will undergo a behavioural questionnaire, and anal swabs which will be tested for HPV and cytology. An HRA will also be performed on all men. Blood will be collected for HIV testing for HIV negative participants, syphilis and storage. Participants will be followed up for three years with one six-monthly visit in the first year then annually. A 6th study visit to discuss all study results will take place 2-3 months after the 5th study visit. A behavioural questionnaire, an anal swab, and HRA will be administered at all follow up interviews.
  Interventions: Procedure: Participants asked questions about recent experiences of anal intercourse in the last six months.; Procedure: High Resolution Anoscopy
- HIV negative homosexual men (Other): Therefore, it is proposed we conduct a longitudinal study of the epidemiology of low risk and high risk HPV infection and related low grade and high grade anal cancers in HIV negative and HIV positive homosexual men who are 35 years or older. Participants are asked questions about recent experiences of anal intercourse in the last six months.
  At baseline, all men (both HIV positive and HIV negative)will undergo a behavioural questionnaire, and anal swabs which will be tested for HPV and cytology. An HRA will also be performed on all men. Blood will be collected for HIV testing for HIV negative participants, syphilis and storage. Participants will be followed up for three years with one six-monthly visit in the first year then annually. A 6th study visit to discuss all study results will take place 2-3 months after the 5th study visit. A behavioural questionnaire, an anal swab, and HRA will be administered at all follow up interviews.
  Interventions: Procedure: Participants asked questions about recent experiences of anal intercourse in the last six months.; Procedure: High Resolution Anoscopy

INTERVENTIONS:
Procedure: Participants asked questions about recent experiences of anal intercourse in the last six months. — Therefore, it is proposed we conduct a longitudinal study of the epidemiology of low risk and high risk HPV infection and related low grade and high grade anal cancers in HIV negative and HIV positive homosexual men who are 35 years or older. Participants are asked questions about recent experiences of anal intercourse in the last six months.
  At baseline, all men (both HIV positive and HIV negative)will undergo a behavioural questionnaire, and anal swabs which will be tested for HPV and cytology. An HRA will also be performed on all men. Blood will be collected for HIV testing for HIV negative participants, syphilis and storage. Participants will be followed up for three years with one six-monthly visit in the first year then annually. A 6th study visit to discuss all study results will take place 2-3 months after the 5th study visit. A behavioural questionnaire, an anal swab, and HRA will be administered at all follow up interviews.
  Other Names: Participants have venepuncture, anal swab and examination under microscope .
Procedure: High Resolution Anoscopy — The HRA is performed on HIV positive and HIV negative participants by study doctor after an examination of the perianal region and perineum. The plastic anoscope is inserted into the anal canal and visualised under high resolution magnification. Biopsy samples will be taken by the clinician for histological assessment if there are any detected abnormalities.
  Other Names: HRA

SUMMARY:
SPANC stands for Study of the Prevention of Anal Cancer. There are more than 100 types of human papillomavirus (HPV). Some HPV types cause genital warts and other types cause more than 90% of anal cancer.

Gay men are over 20 times more likely than others to develop anal cancer.

SPANC is a study of anal (HPV) infection and related anal disease in gay men. The study will provide important information to guide the possible future introduction of anal cancer screening programs for gay men.

DETAILED DESCRIPTION:
Study title: The natural history of anal human papillomavirus (HPV) infection and anal cellular abnormalities in homosexual men.

Protocol version: 7, dated 1 September 2013. Approved by Ethics Committee on 24th October, 2013

Objectives: Among homosexual men aged 35 years or above to determine:

1. Prevalence, incidence and risk factors for specific types of HPV infection.
2. Prevalence, incidence and risk factors for histologically confirmed anal low grade and high grade squamous intraepithelial lesions (LSIL and HSIL).
3. Type-specific rates of clearance and persistence of anal HPV infection.
4. Rates of disease progression, regression and predictors in the spectrum of anal dysplasia.
5. Psychosocial/quality of life impact of anal cytology screening in homosexual men.

Study results will be used to inform possible development of guidelines for carrying out an anal cancer screening program in this population.

The study design is a prospective longitudinal design. Upon enrolment, participants will be followed up for three years to allow the study of both prevalence and incidence of HPV infection and related conditions.

Planned sample size: 600 homosexual men will be screened and enrolled from community based settings in Sydney, Australia.

The inclusion criteria are:

* male homosexual aged 35 years or above;
* HIV positive participants: documented to be HIV positive;
* HIV negative participants: tested HIV negative at recruitment; provision of informed, written consent.

The exclusion criteria are:

* participants unable to attend scheduled follow-up interviews or unwilling to undergo high resolution anoscopies (HRA);
* unable to understand English;
* having bleeding disorders or currently taking anti-anticoagulant medications; *having previously received HRA;
* having ever been diagnosed with anal cancer.

Study procedures:

* At baseline, all men will undergo a behavioural questionnaire, and anal swabs which will be tested for HPV and cytology.
* An HRA will also be performed on all men.
* Blood will be collected for HIV testing for HIV negative participants, syphilis and storage. Participants will be followed up for three years with one six-monthly visits in the first year and then annually. A 6th study visit to discuss all study results will take place 2-3 months after the 5th study visit. A behavioural questionnaire, blood collection (except at six month); an anal swab and HRA will be administered at all follow up interviews.

The SPANC study is a prospective cohort study of the national history of anal human papillomavirus (HPV) infection and anal cellular abnormalities in homosexual men aged 35 years and above in Sydney. It is expected that the study results will be influential in the possible development of an anal cancer screening program in high-risk populations. Data on the natural history of anal HPV infection in homosexual men recruited from community-based settings are rare. We aim to recruit a total of 600 men, 360 HIV-negative and 240 HIV-positive. This will make the SPANC study one of the biggest ongoing anal HPV natural history study in the world to provide critical data on the incidence and clearance of anal HPV infection, progression and regression of pre-cancerous HPV associated anal lesions, the potential psychological impact on men who participate anal cancer screening programs, and the cost-effectiveness of rolling out these programs.

Statistical considerations: Sample size calculation: Assuming the incidence of HSIL is 5 and 15 per cent 100 person-years in HIV negative and HIV positive men, respectively, the 95% confidence intervals will be 4.2-6.0 in the HIV negative arm and 12.6-17.8 per 100 person-years in the HIV positive arm. Analysis plan: HPV prevalence and incidence, including overall, low risk, high risk and individual types, will be calculated according to participant's HIV status. Prevalence and incidence of LSIL and HISL will be calculated in the same fashion. Clearance and persistence of HPV infection, and progression and regression of HSIL will also be determined. Risk factors for prevalent HPV infection and LSIL and HSIL will be analysed using logistical regression. Risk factors for incident conditions will be analysed using Cox regression.

Duration of the study: The study will take place from 13/September/2010 to 21/Dec/2018. Participants will be recruited from 2010 to 2015 and followed up for three years.

ELIGIBILITY:
Inclusion Criteria: Male homosexual aged 35 years or above; HIV positive participants: documented to be HIV positive; HIV negative participants: tested HIV negative at recruitment; provision of informed, written consent.

-

Exclusion Criteria: participants unable to attend scheduled follow-up interviews or unwilling to undergo high resolution anoscopies (HRA); unable to understand English; having bleeding disorders or currently taking anti-coagulant medications; having previously received HRA; having ever been diagnosed with anal cancer.

-

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2010-09-10 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
A natural history study to inform the potential usefulness of a cytology/HPV/HRA based screening program | 3 year cohort study
  Aims to determine the prevalence, incidence and risk factors for type-specific HPV (37 types)

SECONDARY OUTCOMES:
Prevalence, incidence and risk factors for LSIL and HSIL | 3 year cohort study
  To determine if HPV is associated with LSIL and HSIL

CONTACTS AND LOCATIONS:
Overall Officials: Carmella Law, MBBS; FAChSHM;, Principal Investigator — Appplied Medical Research, the Clinical Research Program at St. Vincent's Hospital; David Templeton, MBChB; PhD;, Principal Investigator — RPA Sexual Health, Royal Prince Alfred Hospital
Locations (2):
- Australia (2):
  - Applied Medical Research (AMR CRP), St. Vincent's Hospital, Sydney, New South Wales
  - RPA Sexual Health, Royal Prince Alfred Hospital, Camperdown, Sydney, New South Wales

REFERENCES:
- [Background] Machalek DA, Grulich AE, Hillman RJ, Jin F, Templeton DJ, Tabrizi SN, Garland SM, Prestage G, McCaffery K, Howard K, Tong W, Fairley CK, Roberts J, Farnsworth A, Poynten IM; SPANC Study Team. The Study of the Prevention of Anal Cancer (SPANC): design and methods of a three-year prospective cohort study. BMC Public Health. 2013 Oct 9;13:946. doi: 10.1186/1471-2458-13-946. PMID 24107134
- [Derived] Tong WW, Shepherd K, Garland S, Meagher A, Templeton DJ, Fairley CK, Jin F, Poynten IM, Zaunders J, Hillman RJ, Grulich AE, Kelleher AD, Carr A; Study of the Prevention of Anal Cancer (SPANC) team. Human papillomavirus 16-specific T-cell responses and spontaneous regression of anal high-grade squamous intraepithelial lesions. J Infect Dis. 2015 Feb 1;211(3):405-15. doi: 10.1093/infdis/jiu461. Epub 2014 Aug 19. PMID 25139018
- See also: http://www.nchersurveys.unsw.edu.au/spanc — http://www.kirby.unsw.edu.au